CLINICAL TRIAL: NCT04341532
Title: Bacterial Gene Profiling to Predict Antibiotic Resistance During Cystic Fibrosis Pulmonary Exacerbations
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Jewish Health (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: SAAVED19A0
Record Dates: First submitted 2020-04-02; First posted 2020-04-10 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary exacerbations (PEx) are key events that lead to a decline in health status among CF patients, with many never recovering to baseline health. With the advancement of new CFTR modulators and other therapies increasing the lifespan of those living with CF, it will become increasingly important to have better strategies to manage PEx in order to have better outcomes following treatment. PEx treatment decisions will need to take into consideration the increasing frequency of antimicrobial resistance bacteria and the need to treat multiple types of bacteria at once. The purpose of this study is to analyze sputum samples from CF subjects at the time of PEx in order to identify markers of antimicrobial resistant bacteria and see how those relate to treatment responses. CF patients will be recruited from patients followed by the Adult CF Program at National Jewish Health. Within 48 hours of admission to the hospital for treatment of a PEx, subjects will be enrolled and sputum will be collected. The sputum will be processed and analyzed for the presence of antimicrobial resistant bacteria. These results will be compared to clinical data, such as spirometry and frequency of hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* CF patients 18 years or older who are hospitalized for IV treatment of an acute PEx
* Chronically infected with Pseudomonas aeruginosa and/or Staphylococcus aureus
* Can produce sputum
* Can provide written consent
* Willing to comply with study procedure

Exclusion Criteria:

* Subjects who are not colonized with Pseudomonas aeruginosa and/or Staphylococcus aureus
* The presence of a condition or abnormality that, in the opinion of the Principal Investigator, would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An eligible subject will be a current patient of the Colorado Adult CF Clinic who is being hospitalized at the onset of IV treatment for a pulmonary exacerbation, as diagnosed by a clinic physician, and who is chronically infected with Pseudomonas aeruginosa and/or Staphylococcus aureus.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Targeted amplicon sequencing of sputum | Within 48 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation
  Results from CF specific amplicon panel; this may include number and identity of bacterial species, presence or absence of AMR genes, frequencies of strain types, and AMR genes per total bacteria
Sputum microbiology | Within 48 hours of initiation of IV antibiotic treatment for CF pulmonary exacerbation
  Traditional sputum microbiology results; this may include quantitative culture data for each pathogen, antimicrobial susceptibilities, and minimum inhibitory concentration (MIC)
Change in lung function | At initiation of IV antibiotic treatment and after one week of IV antibiotic treatment
  Change in lung function as measured by FEV1, % predicted.

SECONDARY OUTCOMES:
Changes in hospitalizations | 12 months prior to enrollment to 12 months after enrollment
  Changes in frequency/number of hospitalizations for treatment of CF pulmonary exacerbation
Antimicrobial regimens | Throughout course of hospitalization, on average 14 days
  Type/total number of IV antibiotic doses delivered

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No